CLINICAL TRIAL: NCT05192863
Title: Complete Remission in Patients With Moderately to Severely Active Crohn's Disease Treated With Vedolizumab - A Multicenter, Prospective Observational Cohort Study in Canada, Italy, and Israel
Brief Title: A Study of Vedolizumab in Adults With Crohn's Disease (CD)
Acronym: SUNRISE
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-4038
Record Dates: First submitted 2022-01-11; First posted 2022-01-14 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Crohn's Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with CD: Participants diagnosed with moderately to severely active CD who are initiating vedolizumab intravenous (IV) induction treatment with the option to switch to vedolizumab subcutaneous (SC) treatment, as maintenance therapy in accordance with the current SmPC will be observed prospectively for 18 months.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The main aim of this study is to see if adults with CD treated with vedolizumab have less symptoms and inflammation of the bowel assessed by ultrasonography.

Participants will be treated with vedolizumab according to their clinic's standard practice.

DETAILED DESCRIPTION:
This is a non-interventional, prospective study of participants with moderately to severely active CD who are initiating treatment with vedolizumab according to the current summary of product characteristics (SmPC) in the real world setting.

The study will enroll approximately 100 participants. The data will be collected prospectively at the study sites and will be recorded into electronic case report forms (e-CRFs). All the participants will be assigned to a single observational cohort:

Participants with CD

This multi-center study will be conducted in Canada, Italy, and Israel at specialized gastroenterology centers. The overall duration of the study will be 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Has moderately to severely active CD with a BWT of >3 mm, based on IUS performed within the previous 4 weeks from baseline.
2. Newly initiating IV vedolizumab induction treatment in accordance with the current SmPC either at enrolment or within 2 weeks after enrolment (switch to SC is acceptable at maintenance treatment stage).

Exclusion Criteria:

1. Prior history of intolerability, hypersensitivity to the active substance or to any of the excipients of vedolizumab.
2. Active severe infections such as tuberculosis (TB), sepsis, cytomegalovirus, listeriosis, and opportunistic infections such as Progressive Multifocal Leukoencephalopathy (PML).
3. Cognitive incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
4. Current or previous participation in an interventional clinical trial for CD within the past 30 days, or planned to be enrolled in an interventional clinical trial for CD.
5. Ongoing or planned pregnancy or breastfeeding participants.
6. Active perforating complications or significant current strictures (assessed by IUS, with or without pre-stenotic dilatation) as per clinical judgement.
7. Characteristics precluding IUS visualization of affected bowel segments or normal BWT of <=3 mm for all segments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with moderately to severely active CD initiating vedolizumab therapy in a routine clinical care, with a BWT of >3 mm, based on IUS assessment.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieve Complete Remission 12 Months After Initiation of Vedolizumab Therapy | Baseline up to 12 months
  Complete remission will be measured by corticosteroid-free clinical, biochemical and transmural remission.Corticosteroid-free defined as no usage of any systemic or locally acting steroid.Corticosteroid-free clinical remission defined as Harvey Bradshaw Index (HBI) less than (<) 5 points and no concomitant corticosteroids.HBI score measures disease activity of CD. Clinical parameters:general well-being (0-4,higher score lower well being),abdominal pain(0-3,higher score more severe pain),number of liquid stools/day, abdominal mass (0-3),higher score presence of swelling in abdomen),complications (score 1/item).Total is sum of individual parameters.Score:minimum 0-no pre-specified maximum score,depends on number of liquid stools, higher scores indicating more severe disease.Biochemical remission defined as C-reactive protein(CRP) and fecal calprotectin (FCal) normalization.Transmural remission defined as bowel wall thickness(BWT) of <3 millimeter (mm) for all bowel segments upon IUS.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve Complete Remission | Up to Month 18
  Complete remission will be measured by corticosteroid-free clinical, biochemical and transmural remission. Corticosteroid-free defined as no usage of any systemic or locally acting steroid. Corticosteroid-free clinical remission defined as HBI <5 points and no concomitant corticosteroids. HBI score is used to measure disease activity of CD. Biochemical remission defined as CRP and FCal normalization. Transmural remission defined as BWT of <3 mm for all bowel segments upon Intestinal Ultrasonography (IUS).
Percentage of Participants Who Achieve Corticosteroid-free Clinical Remission | Up to Month 18
  Corticosteroid-free defined as no usage of any systemic or locally acting steroid. Corticosteroid-free clinical remission defined as HBI <5 points and no concomitant corticosteroids. HBI score is used to measure disease activity of CD.
Percentage of Participants Who Achieve Biochemical Remission | Up to Month 18
  Biochemical remission defined as CRP and FCal normalization.
Percentage of Participants Who Achieve Transmural Remission | Up to Month 18
  Transmural remission defined as BWT of <3 mm for all bowel segments upon IUS.
Percentage of Participants Who Achieve Clinical Response | Up to Month 18
  Clinical response is defined as a reduction of greater than or equal to (>=) 3 points from the baseline HBI score. HBI score is used to measure the disease activity of CD.
Percentage of Participants Who Achieve Transmural Response | Up to Month 18
  Transmural response is defined as a minimum reduction of 25 percent (%) of BWT from baseline or absolute BWT less than or equal to (<=) 3 mm upon IUS.
Percentage of Participants With Change, and Reason for Change in Vedolizumab Dosing Frequency | Up to Month 18
Percentage of Participants Who Switched to Vedolizumab SC Formulation | Up to Month 18
Percentage of Participants Who Discontinued Vedolizumab Treatment and Reason for Discontinuation | Up to Month 18
Percentage of Participants With Prior Treatments for CD, and Reason for Discontinuation | Up to Month 18
Percentage of Participants With Concomitant Therapies for CD | Up to Month 18
  Concomitant therapies for CD including introduction and discontinuation of systemic steroids; any changes and reasons for changing including dosing regimen changes, discontinuation, initiation etc.
Percentage of Participants Who Switched to Other CD Therapy After Vedolizumab Discontinuation | Up to Month 18
Percentage of Participants With Acceptance of IUS Monitoring and Assessment | Up to Month 18
  IUS is a 6 item questionnaire visual analogue scale (VAS). Out of 6 items, 2 items has score range 1 (completely unacceptable) to 10 (completely acceptable): Item 1-Acceptability as monitoring tool in IBD; and Item 2-Acceptability of other monitoring tools in IBD including 6 sub items with score range 1 to 10. Item 3- IUS examination leading to improvement of knowledge of their illness with score range 1 (totally useless) to 10 (very useful). Item 4: Tolerability of IUS with score range 1 (no discomfort) to 10 (much discomfort). Item 5: Choice of monitoring modality with score range 1 (most preferred) to 5 (least preferred). Item 6: IUS examination leading to improvement of knowledge/understanding of illness including 5 sub-items with score range of 1 (completely disagree) to 10 (strongly agree). Responses to these 6 questions will be summed to maximum score of 145. The total score range represents participant's experience of IUS and their acceptability to this assessment.
Percentage of Participants With Improved Quality of Life Based on Health-related Quality of Life (HRQoL) as Measured by Short Inflammatory Bowel Disease Questionnaire (SIBDQ) | Baseline up to Month 18
  The SIBDQ is an instrument used to assess quality of life and is a disease-specific HRQoL questionnaire, that consists of 10 questions grouped into four different dimensions: social, bowel, emotional, and systemic, each question is scored on a scale from 1 (a severe problem) to 7 (not a problem at all). The total score will be reported and will range from 10 to 70 with a higher score indicates a better health-related QoL.
Percentage of Participants With CD-related hospitalizations, CD-related emergency room (ER) visits, CD-related surgeries, CD-related flares requiring IV Induction Therapy or IV Corticosteroid Therapy | Up to Month 18
  Health Care Resources Utilization (HCRU) will be calculated as available in the medical record and captured in the eCRF.
Number of Participants Reporting one or More Adverse Drug Reactions (ADRs) | Up to Month 18
Number of Participants Reporting one or More Serious Adverse Events (SAEs) | Up to Month 18
Number of Participants Reporting one or More Adverse Events of Special Interest (AESIs) | Up to Month 18

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Saskatchewan, Saskatoon, Saskatchewan
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Italy (5):
  - Ospedale ASST Rhodense, Rho, Milano
  - Fondazione Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - ASST Fatebenefratelli Sacco, Milan
  - A.O.U. Federico II, Napoli

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language. — https://clinicaltrials.takeda.com/study-detail/3dbbe12c654e4abf?idFilter=%5B%22Vedolizumab-4038%22%5D